CLINICAL TRIAL: NCT02793739
Title: A Pilot Study Examining the Efficacy of Hyaluronic Acid Filler to Correct Volume Loss in the Dorsal Fingers
Brief Title: Hyaluronic Acid Filler for Dorsal Finger Volume Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmur Medical (Other)
Responsible Party: Principal Investigator, Ellen Marmur, MD, Director Marmur Medical, Associate Clinical Professor of Dermatology, Associate Clinical Professor of Genomics and Genetic Science, The Mount Sinai Hospital, Marmur Medical
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GALD2016-01
Record Dates: First submitted 2016-05-19; First posted 2016-06-08 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Personal Satisfaction
Keywords: Safety; Efficacy; Longevity
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 20 subjects (Experimental): 20 subjects will be enrolled to take part in this study and followed for a period of 12 months. Subjects will receive hyaluronic acid filler injection in the dorsal fingers (2-4 syringes) at the initial visit for volume restoration. If warranted, subjects will receive touch-up of hyaluronic acid at day 14 (1-2 syringes). The investigators expect volume restoration to last 9-12 months.
  Interventions: Procedure: Hyaluronic acid filler injection

INTERVENTIONS:
Procedure: Hyaluronic acid filler injection — Hyaluronic acid filler will be injected into the dorsal fingers at day 0 and at day 14 if a touch-up is necessary.

SUMMARY:
Fingers are a part of the body that are often subject to increased signs of aging due to physical use, trauma and exposure to the environment. The FDA's recent approval of a dermal filler, calcium hydroxylapatite, in hands has led to increased patient demand for hand fillers which, in turn, has led to the question of rejuvenation of the dorsal fingers. Due to the different anatomy of the fingers than the dorsal hand plus the new demand to improve the entire hand plus the finger area, we aim to characterize the best approach. Youthful fingers are devoid of wrinkles and often have fuller contours thus hiding the "knuckles" (proximal and distal interphalangeal joints). With aging and loss of subcutaneous tissue volume, fingers become wrinkled, look more skeletal, almost emaciated, and joints become much more prominent, all aesthetic features often disliked by patients. By augmenting the volume in the dorsal fingers, it is possible that the visibility of such bony structures will be decreased, wrinkles will become smoother, and a more youthful appearance of the fingers will be restored.

There have been no published reports, to these investigators' knowledge, of the use of injectable filler into the dorsal fingers for three-dimensional volume correction. The use of exogenous hyaluronic acid (HA) filler in the fingers would be off-label. Given that HA filler has been used safely and effectively in many areas of three-dimensional volume restoration throughout the body, the investigators believe the HA filler may be used to effectively and safely correct volume loss in the fingers. The investigators hope that this study will present current, state of the art, never before reported technique, safety, efficacy and patient satisfaction of HA filler in this region.

DETAILED DESCRIPTION:
At Marmur Medical, subjects will be recruited and consented prior to any study evaluations or procedures; if subjects meet the inclusion/exclusion criteria, participants will be enrolled into this study. Informed consent will clearly say the use of hyaluronic acid filler for the treatment of dorsal finger volume loss is investigational. Subjects will also be compensated for their visits (initial and six follow-ups totalling seven visits). Pre and post treatment photographs will be taken. Subjects will be given lidocaine cream to apply to the area of injection for temporary numbing effect prior to injection (10-15 minutes). Ice packs will also be applied to the area temporarily for numbing effect just prior to injection. The patient's fingers will be injected with 0.5-2.0 mL of hyaluronic acid total at the level of the sub-dermal plane. The injected filler will be molded as needed to optimize the correction of the fingers. Syringes used and amount injected into each finger, as well as the total per hand, will be documented to the 0.1 mL increment (e.g. 3.4 mL). The expected volume needed is 1-2 syringes per subject initially. On Day 14, subjects will return for evaluation and possible touch-up of injectable hyaluronic acid filler if needed (at the injector's discretion). The expected volume needed may be 1-2 syringes per subject for touch-up.

The subjects will return for follow-up at all time-points as follows: day 14 (+/- touch-up hyaluronic acid injection if necessary), 6 weeks, 3/6/9/12 months. The patient and investigator(s) will assess the volume enhancement in the fingers. Subjects will be asked to rate their level of satisfaction with the treatment at follow-up visits (Global Satisfaction Assessment, Natural Look/Feel Scale). In addition, at the initial visit, subjects will be given a 30 day diary to fill out that will evaluate for symptomology after injection (pain, bruising, swelling, redness, sensitivity/tenderness, itching, lumps/bump development, temporary numbness, signs of vascular compromise or other/open comment box). The subject diary will be collected at the 3 month follow-up visit. Statistical analysis of the data gathered will be performed by an outside statistician using tests such as Wilcoxian signed-rank test (for two observations) or Friedman's test (for more than 2 observations) using STAT, version 13. All adverse events will be recorded at every follow-up visit. These events include: redness, swelling, tenderness, nodule development under the skin and restricted range of motion. More serious adverse events include: compartment syndrome, infection at injection site, Tyndall effect, persistent granulomatous change, injection necrosis, persistent erythema with edema, and vascular occlusion causing symptoms such as pain, numbness and necrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Exhibit volume loss and/or increased laxity and wrinkling of the dorsal fingers as determined by the investigator (moderate to severe volume loss).
2. 18 years of age or older at time of consent. May be male or female.
3. Can be of any Fitzpatrick Skin Type (I-VI).
4. Able and willing to give written informed consent and to comply with requirements of this study protocol. The consent form has been standardized in English. For those patients who do not read and understand English, a consent form will be standardized and provided in a language that they read and understand, if possible.

Exclusion Criteria:

1. Children and adolescents (less than 18 years old)
2. Subjects who are not willing or able to prove written consent.
3. Individuals with any significant medical history including skin disorders and eating disorders.
4. Subjects with previous and/or known hypersensitivity to lidocaine, hyaluronic acid, or any of their

   preservatives, wasp/bee/hornet stings, and/or hyaluronidase.
5. Subjects on any substances affecting blood coagulation (i.e. aspirin and other non-steroidal anti-

   inflammatory drugs, warfarin, vitamin E, heparin).
6. Subjects with known blood coagulopathies.
7. Subjects with a compromise of local blood supply (i.e. recent surgery, severe scarring).
8. Subjects with previous history of rheumatologic or collagen vascular disease.
9. Subjects who have received semi-permanent or temporary filler in the fingers in the past 18

   months.
10. Subjects with any history of permanent filler in the fingers.
11. Subjects with dorsal finger volume loss too severe to be treated in one treatment session.
12. Female patients who are planning a pregnancy, currently pregnant or nursing.
13. Failure to sign photographic consent forms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of three-dimensional volume restoration in the dorsal fingers by hyaluronic acid filler using a 5 point volume loss scale | Baseline, Day 14, 6 weeks, 3 months, 6 months, 9 months and 12 months
  At each study visit, the investigator or sub-investigator will collect data regarding efficacy of volume restoration in the dorsal fingers by assessing qualitative changes in volume of the dorsal fingers.

SECONDARY OUTCOMES:
Patient Satisfaction based on the Global Aesthetic Assessment Scale | Day 14, 6 weeks, 3 months, 6 months, 9 months and 12 months
  At each study visit, the participants will fill out surveys regarding global aesthetic improvement (a 7 point scale).
Patient Satisfaction based on the Natural Look/Feel Scale | Day 14, 6 weeks, 3 months, 6 months, 9 months and 12 months
  At each study visit, the participants will fill out surveys regarding natural look/feel of the the product on a 10 point scale.
Patient Satisfaction based on the Subjective Patient Diary | 1 month
  Over the period of 1 month, patients will be documenting subjective pain, tenderness, redness, itching, development of nodules on a scale of 10.
Patients with treatment-related adverse events as reported by patients and confirmed by investigator and/or sub-investigator | Baseline, Day 14, 6 weeks, 3 months, 6 months, 9 months and 12 months
  At each study visits, the investigator or sub-investigator will collect data regarding adverse events occurring after hyaluronic acid filler injection into the dorsal fingers. If participants have concerns regarding adverse events they are encouraged to call the office and see the investigator and/or sub-investigator immediately to discuss these concerns.
Longevity of hyaluronic acid filler in three-dimensional volume restoration of the dorsal fingers | Baseline, Day 14, 6 weeks, 3 months, 6 months, 9 months and 12 months
  Over a period of 12 months, the investigator, sub-investigator and participants will be filling out a singular survey at each visit that will determine how long volume restoration lasts before effects are mitigated by hyaluronic acid filler dissolution.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Marmur, MD, Principal Investigator — Marmur Medical
Locations (1):
- Marmur Medical, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators plan to present data at dermatologic meetings and publish in dermatologic journals. The investigators do not plan to presents individual participant data.